CLINICAL TRIAL: NCT03517358
Title: Virological Suppression in HIV Positive Patients Involved in a Novel, Standardized Adherence Protocol
Brief Title: Virological Suppression in HIV Positive Patients Involved in a Novel Standardized Adherence Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1150661
Record Dates: First submitted 2018-04-10; First posted 2018-05-07 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacy (Active Comparator): service of care: pharmacy
  Interventions: Other: Service of care
- Case management (Active Comparator): service of care: case management
  Interventions: Other: Service of care

INTERVENTIONS:
Other: Service of care — Subjects will be receiving care from case management or clinical pharmacy.

SUMMARY:
This study will look at virologically suppression of patients with HIV who receive pharmacist or case management care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a baseline viral load > 200 copies/ml
* Patients who agree to program enrollment
* Patients ≥ 18 years of age

Exclusion Criteria:

* Pregnant women
* Adults unable to consent
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Percentage of virological suppression | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- One Community Health, Sacramento, California, United States